CLINICAL TRIAL: NCT00910598
Title: A Multicenter Longitudinal Cross-sectional Pilot Study, to Compare RNFL Thickness Measured by OCT After Treatment With Glatiramer or After no Treatment in Patients With CIS With or Without Optic Neuritis or With Early RRMS
Brief Title: Optical Coherence Tomography: Glatiramer in Clinically Isolated Syndrome or Early Relapsing Remitting Multiple Sclerosis (MS)
Acronym: OCTIMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Collaborators: Sanofi (Industry); TEVA Pharmachemie (Unknown)
Responsible Party: E.C.A.M. Sanders, Amphia Ziekenhuis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCT
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Multiple Sclerosis
Keywords: clinically isolated syndrome; relapsing remitting multiple sclerosis; glatiramer acetate; Optical Coherence Tomography
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- glatiramer acetate (Experimental): glatiramer acetate 20 mg s.c. daily for 1 year
  Interventions: Drug: glatiramer acetate
- no treatment (No Intervention): No disease modifying treatment allowed

INTERVENTIONS:
Drug: glatiramer acetate — 20 mg daily s.c. for 1 year
  Other Names: Copaxone
  Arms: glatiramer acetate

SUMMARY:
This is a study in patients with clinically isolated syndrome (CIS) and early relapsing remitting multiple sclerosis (RRMS) to assess the effects of glatiramer acetate (GA) subcutaneously on the condition of the optical nerve in comparison to no medicinal therapy during 12 months and to assess the use of Optical Coherence tomography (OCT), a non-invasive ophthalmological technique, in daily practice as an alternative to magnetic resonance imaging (MRI) scanning for follow-up of these patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a progressive and demyelinating disease of the central nervous system characterized by inflammation and neurodegeneration. It is characterized by an ongoing process of demyelination and axonal loss, even at the beginning of the disease course, which will result in brain atrophy. A first manifestation of clinical definite MS, is called a clinically isolated syndrome (CIS). Brain atrophy occurs even in patients with a CIS. Optic neuritis (ON) is a common feature of a CIS. The axons in the retina represent the most proximal part of the optic nerve which is devoid of myelin. Because the retina is part of the central nervous system (CNS), measurement of the Retinal Nerve Fiber Layer (RFLN) by Optical Coherence Tomography (OCT) offers the opportunity to visualize the unmyelinated axons of the CNS directly. OCT is a non-invasive method to measure the thickness of the optical layer. The thickness of the RNFL is reduced in MS patients with or without ON history.

Glatiramer acetate (GA), an immunomodulatory drug for RRMS and CIS, reduces brain atrophy and stimulates the production of brain-derived neurotrophic factor, which in turn could stimulate neuroregeneration.

In this pilot study we would like to assess the feasibility of OCT measurement in patient with CIS other than ON in the Dutch clinical setting and to assess the effect of GA on the RNFL and visual function in patients with CIS or in early relapsing remitting MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 55 years
* Early relapsing remitting MS, defined as a disease course less than 3 years
* clinically isolated syndrome , defined as optic neuritis (ON) or other than ON
* Currently treated with glatiramer (GA) or currently not treated for MS
* Expanded disability status scale (EDSS) score 0-5
* Able and willing to provide written informed consent prior to enrolment
* Willing and able to comply with the protocol requirements for the duration of the study

Exclusion Criteria:

* Clinical definite multiple sclerosis with a disease course more than 3 years
* Primary progressive multiple sclerosis
* Secondary progressive multiple sclerosis
* Current use of any approved or investigational disease modifying agents for the treatment of MS other than GA.
* Neuromyelitis Optica (Devic's disease)
* Any condition that may interfere with the quality of the OCT scan: clouding of the media, i.e. cataract, pupil which are hard to dilate.
* Contra-indications for Copaxone ® as defined in the Summary of Product Characteristics (SPC) text
* Hypersensitivity to GA or mannitol
* Subject's inability to complete the study or if the subject is considered by the investigator to be for any reason, an unsuitable candidate for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of OCT measurement in patient with CIS with or without optic neuritis or with early RRMS in the Dutch clinical setting | 1 year

SECONDARY OUTCOMES:
Mean change in RNFL in both eyes determined by OCT at baseline, month 3, month 6, month 9, month 12 | 1 year
Other ophthalmological parameters | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: E.C.A.M. Sanders, MD, Study Chair — Amphia ziekenhuis
Locations (2):
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Maasland Ziekenhuis, Sittard

REFERENCES:
- See also: Amphia Hospital Breda Netherlands — http://www.amphia.nl